CLINICAL TRIAL: NCT06134050
Title: Finding the Optimal Aim of Correction in Opening Wedge High Tibial Osteotomy Using 3D Printed Patient-specific Instrumentation (PSI). An RCT Comparing Correction Aimed at 62% Versus 55%.
Brief Title: Finding the Optimal Aim of Correction in Opening Wedge High Tibial Osteotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Oslo University Hospital (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS001
Record Dates: First submitted 2023-06-23; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis, Knee; Knee Pain Chronic; Arthralgia
Keywords: osteotomy; knee; osteoarthritis; 3D print; PSI; High tibial osteotomy; Knee overload; Inertial measurement units; IMU; wearable sensors; gait analysis; accelerometer
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants blinded. Care provider/surgeon not possible to mask. Investigator masked. Outcome assessor masked/blinded data set.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 55% correction (Experimental): HTO using PSI targeted at 55% correction axis
  Interventions: Procedure: Procedure: HTO using PSI aiming at 55% correction
- 62% correction (Active Comparator): HTO using PSI targeted at 62% correction axis
  Interventions: Procedure: Procedure: HTO using PSI aiming at 62% correction

INTERVENTIONS:
Procedure: Procedure: HTO using PSI aiming at 55% correction — HTO using PSI designed to achieve correction to 55% tibial width.
  Arms: 55% correction
Procedure: Procedure: HTO using PSI aiming at 62% correction — HTO using PSI designed to achieve correction to 62% tibial width.
  Arms: 62% correction

SUMMARY:
The purpose of this RCT is to investigate whether high tibial osteotomy using 3D printed patient specific guides aiming at 55% correction is non-inferior to aiming at 62%.

DETAILED DESCRIPTION:
HTO should play a major role in modern treatment algorithms for knee overload and osteoarthritis. By transferring load from the failing/osteoarthritic compartment of the knee to a healthier compartment, HTO can delay or stop the progression of osteoarthritis at an early stage. This can remove pain and increase knee function, making return to work, activities and sport possible. HTO may delay or avoid the need for total knee replacement for >10 years for at least 80% of patients.

The optimal target for the postoperative mechanical axis of the leg is not yet clarified. Both under- and overcorrection can lead to unfavourable results. The classical Fusjisawa´s point of 62%, or approximately 3 deg. of valgus, is still often used as the optimal target, and studies show good clinical results and longevity. With an often accepted accuracy of +/- 3 deg. with conventional methods, the accepted postoperative range of valgus will be from 0 deg. to 6 deg. But the optimal range is possibly much narrower. Recent studies suggest a narrower range and less overcorrection.

3D-printed patient specific instrumentation (PSI) is based on CT of the individual patient´s knee, data simulation of the planned correction and subsequent 3D printed guides for each patient. The PSI design varies, but involves a positioning guide fitting only in position one the proximal tibia, a cutting guidance and a wedge opening guide. PSI seem to improve accuracy to the level of approximately +/- 1 deg. from the preplanned correction and leads to fewer unacceptable outliers compared to the conventional methods available. Improved accuracy has not shown to yield better clinical results.

In the future the target axis should possibly be individualized, based on the pathology treated, gait analyses and data simulations.

Modern gait analysis using wearable accelerator sensors, often referred to as inertial measurement units (IMUs) is rapidly evolving. By coupling individualized and accurate osteotomy with gait analysis using wearable sensors, one could better predict and understand how to normalise each individual patients´ gait pattern and possibly improve patient satisfaction and function after surgery.

By coupling the highly accurate PSI method, an angular stable implant and a composite of outcomes based on radiology, validated patient reported outcome measures and gait analysis, our RCT can investigate if a correction target of 55% is non-inferior to the common 62%.

The study will be designed as a continuous outcome non-inferiority trial where KOOS QoL subscale is used as the primary outcome and the basis for sample size calculation. The Minimal Clinical Important Difference (MCID) for KOOS QoL regarding HTO is 16.5 points. A presumed standard deviation (SD) of 23 points is obtained from a previous study on a similar population. A one-sided t-test power analysis with 2.5% significance level and 80% power level indicates that 31 patients would be needed in each group. In total 70 patients is planned to be included, which takes into account up to 10% dropout rate and some uncertainty regarding the predicted score values.

Statistics:

The primary outcome will be analyzed with a linear mixed model, where the measurements from all time points will be included. The main effect measure will be the between-group difference in change from baseline to two years, which will be estimated with a 95% confidence interval and a P-value for non-inferiority where the null hypothesis is that osteotomy correction to the 55% target is inferior to the correction to the 62% target and the alternative states that it is not. Inferiority is determined by KOOS QOL difference of at least MCID.

Paired samples t-tests will be used to analyze differences between pre- and postoperative measurements on X-rays within each group. Independent samples t-tests will be used to analyze differences between groups. A p-value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients having accepted and signed the informed consent form before surgery
* Patients aged 30-60 years
* Patients with an indication for primary HTO based on anamnestic, clinical and radiological findings leading to the diagnosis of major medial knee compartment overload symptoms
* Mechanical varus axis of 3-9 deg. (calculated on full length weightbearing X-ray (FLWB))
* Correctable angular deformity on the tibia only (medial proximal tibial angle (MPTA) + planned correction < 95 deg. Lateral distal femoral angle (LDFA) <92 deg.)
* Maximal calculated gap height 14 mm
* Only the first knee will be included if later contralateral HTO

Exclusion Criteria:

* Inflammatory arthritis (Rheumatoid Arthritis, Bechterew arthritis, Psoriatic Arthritis)
* Patients using Prednisolone perorally
* Smokers (need to quit preoperatively)
* Significant overweight (Body Mass Index > 35)
* Earlier fractures in affected leg with fracture malalignment >5 deg.
* Extension deficit >10 deg. in the affected knee
* Earlier septic arthritis/osteomyelitis in the affected leg
* Previous major surgery affecting leg function. Earlier knee arthroscopic procedures like ACL-reconstruction are not excluded
* Planned combined procedures involving HTO + ACL/PCL-reconstruction, meniscal transplantation or meniscal root fixation is excluded
* Neurologic disease with symptoms affecting the leg
* Serious illness or other factors that make communication, follow-up or rehabilitation difficult (e.g. alcohol or drug abuse, psychiatric disease, non-Norwegian speakers).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score subscore Quality of Life (KOOS QOL), 0-100, 100 best score | 24 months
  Knee related Quality of Life

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score 12 Short form (KOOS-12), 0-100, 100 best score | 24 months
  Knee related pain, symptoms, ADL, QoL and function
Forgotten Joint Score-12(FJS-12), 0-100, 100 best score | 24 months
  Knee related symptoms and function
EuroQol-5D (EQ-5D), index 0-1, 1 best score | 24 months
  Health related quality of life
University of California at Los Angeles activity level (UCLA), 0-10, 10 most active | 24 months
  Activity level score
Ground contact time (milliseconds) | 24 months
  Accelerometer based gait analysis

OTHER OUTCOMES:
HKA X-ray measures (Standing Hip-Knee-Ankle x-ray) | 6 months
  MPTA/JLCA/LDFA/HKA angles

CONTACTS AND LOCATIONS:
Overall Officials: Tor Kjetil Nerhus, MD, PhD, Principal Investigator — Martina Hansens Hospital

IPD SHARING:
Plan to Share IPD: No